CLINICAL TRIAL: NCT04746352
Title: Effectiveness of Self-myofascial Release Combined With Biofeedback and Electrical Stimulation for the Management of Myofascial Pelvic Pain
Brief Title: Effectiveness of Self-myofascial Release Combined With Biofeedback and Electrical Stimulation for the Management of MFPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Yang Shen, Vice President, Zhongda Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Zhongda Hospital
Record Dates: First submitted 2021-02-01; First posted 2021-02-09 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Myofascial Pelvic Pain
MeSH Terms: interventions — BES

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BES-SMFR group (Experimental): Using the same Vishee neuro-muscle stimulator as the sEMG assessment with a vaginal probe was inserted into the vagina and placed close to the PFMs. Three standardized programs were used in our study: (1) Tens electricity (first program): 5 min of 50-280 Hz frequency and a pulse duration of 50 µs. (b) Endorphin electricity (second program): 5 min of 1-10 Hz frequency and a pulse duration of 200 µs. (c) Spasmolysis electricity (third program): 5 min of 1-2 Hz frequency and a pulse duration of 300 µs. At the same time, patients could learn about their neuromuscular activity through the biofeedback instrument, abdominal breathing for 5 sec was necessary when PFMs were overactive.
  Interventions: Procedure: BES-SMFR
- BES group (Active Comparator): 1. A standardized and structured vaginal examination was performed by digital palpation to identify pelvic floor active MTrPs, and then pain mapping was developed for the patient's use.
  2. Patients were required to participate in intensive training regarding myofascial release techniques. (I) Pressing: press directly on a specific MTrP with gentle, slow pressures (2kg/cm2) using a flat palpation, the pressure was sustained until the participant perceived the pain decreased and taut band released, and then gradually increased to previous level of MTrPs tension and maintained until a reduction of pain again. The process was usually 3 to 5 repetitions for 90 sec. (II) Stretching: stretch in parallel to the direction of the myofascial to facilitate elongation of a contracted muscle. (III) Strumming: stroking and strumming the affected muscles region with the fingertips to aid in MTrPs tension release, the initial pressure was small and increased gradually until the patients adapted.
  Interventions: Procedure: BES

INTERVENTIONS:
Procedure: BES-SMFR — For the BES intervention, it was performed using the same Vishee neuro-muscle stimulator as the sEMG assessment with a vaginal probe was inserted into the vagina and placed close to the PFMs. At the same time, patients could learn about their neuromuscular activity through the biofeedback instrument, abdominal breathing for 5 sec was necessary when PFMs were overactive. BES was performed once every 2 days for 4 weeks.
  Arms: BES-SMFR group
Procedure: BES — First, a standardized and structured vaginal examination was performed by digital palpation to identify pelvic floor active MTrPs, and then pain mapping was developed for the patient's use. Second, patients were required to participate in intensive training regarding myofascial release techniques. Following the training, SMFR was regularly performed by at home for 5 minutes daily for 4 weeks. SMFR was confirmed with patients at all their follow up visits.
  Arms: BES group

SUMMARY:
Myofascial pelvic pain (MFPP) caused by myofascial trigger points (MTrPs) is a major contributor of female chronic pelvic pain. However, the effect of the patient's self-myofascial release (SMFR) is not clear. Current study is to investigate the effect of SMFR combined with biofeedback and electrical stimulation (BES) therapy compared with BES alone in patients with MFPP.

DETAILED DESCRIPTION:
68 patients was enrolled and randomly allocated into two groups: BES-SMFR group (n=34) and BES group (n=34). Every patient received 4 weeks treatment, and was evaluated at baseline (T0), 4-week post-intervention (T4) and 12-week follow-up (T12). The primary outcome was pain intensity. The secondary outcomes were degree in activation of MTrPs, surface electromyography (sEMG) levels, and Patient Global Impression of Improvement (PGI-I).

ELIGIBILITY:
Inclusion Criteria:

1. age between 18 and 70 years;
2. presence of persistent chronic pelvic pain ≥ 4 points on a 10 points numeric rating scale for at least 3 months;
3. at least one active MTrP in one of muscle group including obturator internus, levator ani, piriformis, coccygeus on pelvic examination.

Exclusion Criteria:

1. diseases of the urinary, genital, colorectal systems;
2. prolapse of the pelvic organ;
3. a history of pelvic rehabilitation within the 3 months prior to study;
4. psychiatric disorders;
5. pregnancy;
6. breastfeeding.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
The change of pain intensity | Up to 12 weeks
  Pain intensity was calculated by using the visual numeric rating scale (NRS), which is a 11-point rating scale ranging from "0" (no pain) to "10" (worst pain imaginable) . For each patient, the NRS referred to pain elicited while palpating bilaterally each PFM groups and was averaged pain across all the muscles. Upon palpation, the patient was asked to place in a resting, semi-recumbent position with legs supported by pillow to prevent excessive tension in the PFMs.

SECONDARY OUTCOMES:
The degree in activation of MTrPs | Up to 12 weeks
  MTrPs were considered as active when the following criteria was met: (1) Presence of a palpable taut band in the muscle; (2) Presence of a hypersensitive spot in the taut band; (3) Local twitch response elicited by snapping palpation; (4) Reproduction of the typical referred pain pattern in response to the compression of tender spots; and (5) Spontaneous presence of the typical referred pain pattern. Active MTrPs localized mainly in the bilateral obturator internus, levator ani, piriformis and coccygeus were assessed respectively by pelvic floor manual palpation. Using the inclusion criterion of having active MTrPs at least one in the bilateral muscles as a cutoff point.
Surface electromyography (sEMG) levels of the PFMs | Up to 12 weeks
  The PFMs sEMG assessment was performed based on Glazer protocol by using the device of Vishee neuro-muscle stimulator (MyoTrac Infiniti, model SA9800, Thought Technology Ltd., Montreal, Canada). The sEMG amplitude mean value based on Glazer protocols for selected tasks were follows: 60-s pretest resting baseline, assessing the resting amplitude of PFM before the test sequence; 5 rapid contractions (quick flicks), assessing fast muscles function; 60-s endurance contraction, assessing slow muscles function; 60-s posttest resting baseline, assessing the resting amplitude of PFM after the test sequence.
The score of Patient Global Impression of Improvement (PGI-I) | Up to 12 weeks
  PGI-I is a patient self-reporting evaluation that assesses overall perception of response to treatment according to a 7-point scale, including very much worse, much worse, a little worse, no change, a little better, much better or very much better, with lower scores indicating more favorable outcomes. Better response to treatment was considered when a PGI-I score < 3 (very much better or much better).

CONTACTS AND LOCATIONS:
Overall Officials: Yang Shen, MD,PhD, Study Director — Zhongda Hospital
Locations (1):
- Zhongda Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No